CLINICAL TRIAL: NCT02840916
Title: Laser Acupuncture Therapy in Patients With Postpartum Weight Retention: A Randomized Controlled Trial
Brief Title: Laser Acupuncture for Postpartum Weight Retention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wen-Long Hu, Deputy director, Department of Chinese Medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG8C0691
Record Dates: First submitted 2016-07-14; First posted 2016-07-21 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Postpartum Weight Retention
Keywords: Laser acupuncture; Postpartum weight retention; Obesity
MeSH Terms: conditions — Gestational Weight Gain; Obesity | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- verum laser acupuncture (Experimental): verum laser acupuncture
  Interventions: Procedure: laser acupuncture
- sham laser acupuncture (Sham Comparator): sham laser acupuncture (no laser output)
  Interventions: Procedure: sham laser acupuncture

INTERVENTIONS:
Procedure: laser acupuncture — Subjects were treated at acupoints including the Stomach and Hunger points of the ear, ST25, ST28, ST40, SP15, CV9, and SP6 by using laser acupuncture (GaAlAs laser, maximal power, 150 milliwatt; wavelength, 810 nm; area of probe, 0.03 cm2; power density, 5 W/cm2; pulsed wave; 5.625 J/ cm2) over 5 sessions per week, 12 treatment sessions in total.
  Other Names: low-level laser therapy
  Arms: verum laser acupuncture
Procedure: sham laser acupuncture — Subjects underwent sham laser acupuncture treatment without any laser output. The acupuncture points, application duration, and total number of treatments were similar to those in verum laser acupuncture group.
  Arms: sham laser acupuncture

SUMMARY:
Objective: To determine the therapeutic effect of acupuncture on postpartum weight retention.

Methods: 66 subjects after delivery with postpartum weight retention will be randomly divided into laser acupuncture and control group. A single-blind clinical trial will be conducted and the subjects will be treated with verum or sham laser acupuncture 5 sessions per week. After about 3 weeks of treatment, the differences of the subjects' body weight, body mass index, and waist circumference will be analyzed with ANOVA between laser acupuncture and control group.

DETAILED DESCRIPTION:
Objective: Gestational weight gain and weight retention at 1 year after delivery are associated with long-term obesity. The investigators aimed to investigate the effect of laser acupuncture therapy (LAT) on postpartum weight control.

Methods: The investigators randomly assigned 66 subjects with postpartum weight retention to a laser acupuncture group and control group. The subjects were treated at acupoints including the Stomach and Hunger points of the ear, ST25 (Tianshu), ST28 (Shuidao), ST40 (Fenglong), SP15 (Daheng), CV9 (Shuifen), and SP6 (Sanyinjiao) by using verum or sham laser acupuncture over 5 sessions per week. After 12 treatment sessions, the differences in the body mass index (BMI), body fat percentage (BFP), and waist-to-buttocks ratio (WBR) of the patients were analyzed, and compared between the laser acupuncture and control groups via analysis of variance, chi-square tests, and stepwise regression tests.

ELIGIBILITY:
Inclusion Criteria:

* postpartum duration of <1 month;
* body mass index (BMI) > 25;
* age > 20 years;
* did not use any other medications for weight loss during the study period; and
* provided informed consent.

Exclusion Criteria:

* presence of a pacemaker;
* history of seizure or epilepsy;
* taking immunosuppressant medication;
* cancer;
* infectious disease of the skin;
* taking medications for weight loss, including Chinese herbal preparations, during the study period;
* receiving other treatment, including supplements, herbs, and medications for weight gain prior to entering the study;
* comorbidities (hypothyroidism, renal disease, etc.) that the physician believes would affect the findings;
* unable to undergo LAT due to other medical conditions; and
* lack of informed consent.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hu WL, Chang CH, Hung YC. Clinical observations on laser acupuncture in simple obesity therapy. Am J Chin Med. 2010;38(5):861-7. doi: 10.1142/S0192415X10008305. PMID 20821818

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Verum Laser Acupuncture | Sham Laser Acupuncture
Started | 33 | 33
Completed | 32 | 30
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verum Laser Acupuncture | Sham Laser Acupuncture | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 30 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.88 (4.31) | 35.70 (3.72) | 35.28 (4.02)
Gender [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI)
Description: The BMI was assessed by an evaluator who was blinded to the intervention details from the beginning through study completion, up to 3 weeks, and 3 months after study completion.
Time Frame: up to 3 weeks, 3 months after study completion
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Verum Laser Acupuncture | Sham Laser Acupuncture
Number analyzed (Participants) | 32 | 30
kg/m^2
  baseline | 33.62 (3.19) | 28.03 (3.04)
  up to 3 weeks | 26.90 (2.29) | 26.99 (3.45)
  3 months after study completion | 26.16 (2.40) | 26.64 (3.40)

2. Secondary Outcome: Waist-to-buttock Ratio (WBR)
Description: The WBR was assessed by an evaluator who was blinded to the intervention details from the beginning through study completion, up to 3 weeks.
Time Frame: up to 3 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Verum Laser Acupuncture | Sham Laser Acupuncture
Number analyzed (Participants) | 32 | 30
ratio
  baseline | 0.93 (0.06) | 0.92 (0.06)
  up to 3 weeks | 0.92 (0.05) | 0.90 (0.05)

3. Secondary Outcome: Body Fat Percentage (BFP)
Description: The BFP was assessed by an evaluator who was blinded to the intervention details from the beginning through study completion, up to 3 weeks.
Time Frame: up to 3 weeks
Measure: Mean (Standard Deviation); unit: % of body weight
Arm/Group | Verum Laser Acupuncture | Sham Laser Acupuncture
Number analyzed (Participants) | 32 | 30
% of body weight
  baseline | 36.94 (2.65) | 36.02 (3.87)
  up to 3 weeks | 35.75 (3.05) | 35.37 (3.90)

ADVERSE EVENTS:
Time Frame: 3.75 months
Arm/Group | Verum Laser Acupuncture | Sham Laser Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

LIMITATIONS AND CAVEATS:
The postpartum weight trend cannot be assessed. The average duration of admission in our postpartum care center was 18.6 days. Some confounders should also be considered. The lack of follow-up for BFP and WBR after 1 and 3 months may be limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes